CLINICAL TRIAL: NCT06111924
Title: Effects of Telerehabilitation Versus Clinic-based Task-oriented Circuit Training on Upper Extremity Functions and Quality of Life in Parkinson's Patient.
Brief Title: Effects of Telerehabilitation Versus Clinic-based Task-oriented Circuit Training in Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0042250 Zunaira Ahmad
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Quality of Life; Telerehabilitation; Task oriented circuit training; Upper limb dysfunction
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task oriented circuit training based telerehabilitation (TOCT-TR) group (Experimental): This group will recieve Task oriented circuit training based telerehabilitation (TOCT-TR) via video conference call in 18 sessions.
  Interventions: Other: Task oriented circuit training based telerehabilitation
- Clinic based Task oriented circuit training (TOCT-CR) group (Experimental): This group will recieve In person treatment at clinical setting that will be Task oriented circuit training based telerehabilitation in 18 sessions.
  Interventions: Other: Clinic based Task oriented circuit training

INTERVENTIONS:
Other: Task oriented circuit training based telerehabilitation — Task oriented circuit training based telerehabilitation (TOCT-TR) via video conference call will be provided for 6 weeks, thrice a week in total18 sessions. Total 15 exercises will be performed by patient in a session of 60 minutes. Duration per exercise will be 3 minutes and a rest interval of 1 will be provided after each exercise.
  Arms: Task oriented circuit training based telerehabilitation (TOCT-TR) group
Other: Clinic based Task oriented circuit training — Clinic based Task oriented circuit training (TOCT-CR) will be provided in clinic as in person training for 6 weeks, thrice a week in total18 sessions. Total 15 exercises will be performed by patient in a session of 60 minutes. Duration per exercise will be 3 minutes and a rest interval of 1 will be provided after each exercise.
  Arms: Clinic based Task oriented circuit training (TOCT-CR) group

SUMMARY:
This randomized clinical trial aims to determine effects of Telerehabilitation versus clinic-based task-oriented circuit training on upper extremity functions and quality of life in Parkinson's patient.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder that primarily affects the motor system. It is also affecting dexterity of upper limb. Working on its rehabilitation is important question these days. There is growing evidence that intensity and task-specificity of practice delivered by physical- (PT) may be effective and compliment to pharmacological and surgical treatments. Notably, task specific training improves the patient's abilities in ADL and increases levels of participation. This study aims to compare the effects of telerehabilitation and clinic-based task-oriented circuit training on upper extremity functions and quality of life in Parkinson's patients. Telerehabilitation offers increased accessibility, personalized care, and continuity of therapy. It provides therapy in a convenient way and allows for remote monitoring and feedback.

This randomized clinical trial will be conducted at Lahore general hospital and Sehat Medical complex, Lahore. Diagnosed cases of Parkinson's disease falling in Stage 1 and 2 according to Hoehn-Yahr Classification of Disability Scale with Cognition level according to mini-mental state examination (MMSE) score >24 will be included. Sample will be selected by non-probability convenient sampling technique. Patients will be enrolled and assessed for eligibility criteria. Randomization will be done by sealed envelope method and allocated into two groups, one will get telerehabilitation based task-oriented circuit training TOCT-TR and other group will receive clinic-based task-oriented circuit training TOCT-CR. Patients will be blinded about intervention group. Interventions will be applied for 6 weeks. Pre and post treatment assessment will be done by assessor blinded to study. Thus, it will be double blinded study. Analysis will be done by SPSS 29 version. The findings can contribute to the growing evidence base supporting the use of telerehabilitation in Parkinson's disease management and guide future rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 40-70 years.
* Both gender male and female.
* Diagnosed cases of Parkinson's disease
* Stage 1 and 2 Parkinson's according to Hoehn-Yahr Classification of Disability Scale
* Cognitive stability as defined by a mini-mental state examination (MMSE) score >24.
* Availability of technical instruments for video-call (tablet, laptop, or computer/webcam) and ability to use them by patients and/or caregiver.
* Availability and motivation of patients to participate to a 6-weeks telerehabilitation program

Exclusion Criteria:

* Visual loss
* Hearing loss
* Any musculoskeletal disorder in which exercises are contraindicated. (Trauma, fracture, dislocation or subluxation etc.)
* Secondary neurological, orthopedic, or systemic disorders preventing independent standing and walking.
* Severe peripheral vestibular dysfunction
* Co-morbidity with non-stabilized major medical illnesses.
* Presence of freezing of gait (FOG).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Hoehn-Yahr Classification of Disability Scale | 6th week
  Change from baseline. (For classification of disability) The Hoehn and Yahr Scale is used to measure how Parkinson's symptoms progress and the level of disability. It included stages 1 to 5. Stage 1 defines, Unilateral involvement only usually with minimal or no functional disability and stage include Bilateral or midline involvement without impairment of balance. Patients with these 2 stages will be included in study.
Jebsen Taylor Hand Function test | 6th week
  Change from baseline. (For upper limb function dexterity) The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL). The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, simulated feeding, stacking, and lifting large, lightweight, and heavy objects. Total score is the sum of time taken for each sub-test, which are rounded to the nearest second. Shorter times indicate better performance. JTHFT had moderate to high test-retest reliability and excellent intra rater reliability (r=0.84 and 0.85, P<0.05)
Box and Block Test | 6th week
  Change from baseline. (For manual dexterity) The Box and Block Test (BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test. It can be used with a wide range of populations, including clients with stroke. Clients are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Score each hand separately. Higher scores are indicative of better manual dexterity. Excellent test-retest reliability of the right hand for subjects with impairment (ICC= 0.90) and of the left hand for subjects with impairment (ICC= 0.89)
Parkinson's Disease Questionnaire (PDQ-8) | 6th week
  Change from baseline. (For Quality of life) The 8-item version of the Parkinson's Disease Questionnaire (PDQ-8) is a shortened version of the 39-item Parkinson's Disease Questionnaire (PDQ-39). It was developed to reduce the respondent burden and increase convenience for use among persons with Parkinson's Disease in clinical settings. PDQ-8 was constructed by taking one question from each domain of PDQ-39. To assess quality of life. The PDQ-8 has acceptable internal consistency (Cronbach's α = 0.80; item-scale correlation efficient: 0.56-0.72).

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Salmon R, Preston E, Mahendran N, Ada L, Flynn A. People with mild Parkinson's disease have impaired force production in upper limb muscles: A cross-sectional study. Physiother Res Int. 2023 Jan;28(1):e1976. doi: 10.1002/pri.1976. Epub 2022 Oct 20. PMID 36266769
- [Background] Varalta V, Evangelista E, Righetti A, Morone G, Tamburin S, Picelli A, Fonte C, Tinazzi M, Di Vico IA, Waldner A, Filippetti M, Smania N. Effect of Upper Limb Motor Rehabilitation on Cognition in Parkinson's Disease: An Observational Study. Brain Sci. 2022 Dec 8;12(12):1684. doi: 10.3390/brainsci12121684. PMID 36552144
- [Background] Soke F, Guclu-Gunduz A, Kocer B, Fidan I, Keskinoglu P. Task-oriented circuit training combined with aerobic training improves motor performance and balance in people with Parkinson's Disease. Acta Neurol Belg. 2021 Apr;121(2):535-543. doi: 10.1007/s13760-019-01247-8. Epub 2019 Nov 18. PMID 31741209
- [Background] Vanbellingen T, Nyffeler T, Nigg J, Janssens J, Hoppe J, Nef T, Muri RM, van Wegen EEH, Kwakkel G, Bohlhalter S. Home based training for dexterity in Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2017 Aug;41:92-98. doi: 10.1016/j.parkreldis.2017.05.021. Epub 2017 May 25. PMID 28578819
- [Background] Bianchini E, Onelli C, Morabito C, Alborghetti M, Rinaldi D, Anibaldi P, Marcolongo A, Salvetti M, Pontieri FE. Feasibility, Safety, and Effectiveness of Telerehabilitation in Mild-to-Moderate Parkinson's Disease. Front Neurol. 2022 Jun 16;13:909197. doi: 10.3389/fneur.2022.909197. eCollection 2022. PMID 35785358
- [Background] Eldemir S, Guclu-Gunduz A, Eldemir K, Saygili F, Yilmaz R, Akbostanci MC. The effect of task-oriented circuit training-based telerehabilitation on upper extremity motor functions in patients with Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2023 Apr;109:105334. doi: 10.1016/j.parkreldis.2023.105334. Epub 2023 Feb 28. PMID 36917914
- [Background] Zare M, Ozdemir H, Tavsan MY, Tuna F, Sut N, Guler S, Kabayel DD. Effect of activity-based training versus strengthening exercises on upper extremity functions in Parkinson's patients; A randomized controlled, single blind, superiority trial. Clin Neurol Neurosurg. 2022 Jul;218:107261. doi: 10.1016/j.clineuro.2022.107261. Epub 2022 Apr 29. PMID 35567829
- [Background] Voola SI, Hema S. Effectiveness of tele rehabilitation on manual dexterity and its impact on quality of life in patients with Parkinson's disease: A pilot study. Indian Journal of Physiotherapy & Occupational Therapy Print-(ISSN 0973-5666) and Electronic-(ISSN 0973-5674). 2020;14(2):186-93.
- [Background] Ozkul C, Guclu-Gunduz A, Eldemir K, Apaydin Y, Gulsen C, Yazici G, Soke F, Irkec C. Effect of task-oriented circuit training on motor and cognitive performance in patients with multiple sclerosis: A single-blinded randomized controlled trial. NeuroRehabilitation. 2020;46(3):343-353. doi: 10.3233/NRE-203029. PMID 32310197
- [Background] Cikajlo I, Hukic A, Dolinsek I, Zajc D, Vesel M, Krizmanic T, Blazica B, Biasizzo A, Novak F, Peterlin Potisk K. Can telerehabilitation games lead to functional improvement of upper extremities in individuals with Parkinson's disease? Int J Rehabil Res. 2018 Sep;41(3):230-238. doi: 10.1097/MRR.0000000000000291. PMID 29757774
- [Background] Foki T, Vanbellingen T, Lungu C, Pirker W, Bohlhalter S, Nyffeler T, Kraemmer J, Haubenberger D, Fischmeister FP, Auff E, Hallett M, Beisteiner R. Limb-kinetic apraxia affects activities of daily living in Parkinson's disease: a multi-center study. Eur J Neurol. 2016 Aug;23(8):1301-7. doi: 10.1111/ene.13021. Epub 2016 May 1. PMID 27132653
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Kasten M, Bruggemann N, Schmidt A, Klein C. Validity of the MoCA and MMSE in the detection of MCI and dementia in Parkinson disease. Neurology. 2010 Aug 3;75(5):478; author reply 478-9. doi: 10.1212/WNL.0b013e3181e7948a. No abstract available. PMID 20679642
- [Background] Modestino EJ, Reinhofer A, Blum K, Amenechi C, O'Toole P. Hoehn and Yahr staging of Parkinson's disease in relation to neuropsychological measures. Front Biosci (Landmark Ed). 2018 Mar 1;23(7):1370-1379. doi: 10.2741/4649. PMID 29293439